CLINICAL TRIAL: NCT02376673
Title: A Randomized Controlled Trial Comparing a Children's Book to Brochures for Safe Sleep Education in an At-Risk Population Enrolled in a Home Visitation Program
Brief Title: Comparing Children's Book to Brochures for Safe Sleep Education in a Home Visiting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: de Cavel Family SIDS Foundation (Unknown); Every Child Succeeds (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CincinnatiChildrens
Record Dates: First submitted 2015-02-19; First posted 2015-03-03 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Sudden Infant Death Syndrome (SIDS)
Keywords: Pediatric Health Literacy; Home Literacy Orientation; safe sleep
MeSH Terms: conditions — Sudden Infant Death | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brochures (Active Comparator): Mothers in this arm will receive safe sleep education from home visitors using standard brochures (including 1-page handouts and pamphlets) that are customarily used in this home visiting program.
  Interventions: Other: Standard Brochures
- Children's Book (Experimental): Mothers in this arm will receive safe sleep education from home visitors using a specially-designed children's book incorporating American Academy of Pediatrics safe sleep guidelines.
  Interventions: Other: Children's Book

INTERVENTIONS:
Other: Children's Book — A specially-designed, illustrated (full color) children's book written at a first-grade level, conveying American Academy of Pediatrics safe sleep guidelines through the story. Expanded guidelines are listed on the back cover, at a 4th grade reading level. This book will be exclusively used for safe sleep education at 3 study home visits: prenatal between 32 weeks and term, 1 week postnatal, and 2 months postnatal. The mother will be encouraged to share the book with her baby.
  Other Names: Sleep Baby, Safe and Snug
  Arms: Children's Book
Other: Standard Brochures — An assortment of standard safe sleep educational brochures provided by home visitors during prescribed home visits, covering various recommendations for safe sleep.
  Other Names: What does a safe sleep environment look like?; Bright Futures - Newborn Visit; Home Safe Home - Sleep; Helping Baby Back to Sleep; Sleep and your 1-3 month-old
  Arms: Brochures

SUMMARY:
This randomized controlled trial compares a specially-designed children's book to standard brochures for safe sleep education and reduction of Sudden Infant Death Syndrome (SIDS) risk in a high-risk population of young, first-time mothers enrolled in a home visitation program. Roughly half of the mothers will receive safe sleep education via the book, the other half via brochures, during prescribed home visits. Our study will assess differences in safe sleep knowledge, adherence to recommendations, satisfaction with materials used, and attitudes towards reading with their baby. Our hypothesis is that these will be higher in the group receiving the book, due to simpler language, appealing illustrations, emotional connection, and repeated exposures via shared reading.

DETAILED DESCRIPTION:
Safe sleep and health literacy are priorities at national, state, and local levels. While greatly improved since the launch of the Back to Sleep campaign in the 1990s, the rate of sleep-related infant deaths, notably Sudden Infant Death Syndrome (SIDS), has been stagnant for over a decade. While printed materials are widely distributed for SIDS education, to date none have been proven effective, and overall satisfaction has been low. Reasons include passive delivery, unappealing content, and excessively high reading level, especially for low-socioeconomic status populations. Evidence suggests that an ideal strategy involves printed materials combining simplicity, emotional appeal, cultural sensitivity, and low reading level, conveyed by health care practitioners and reviewed multiple times. Children's books are a potentially ideal medium for this, combining pictures and text to invoke emotion and inspire a shared parent-child experience that is valued and repeated.

This is a randomized controlled trial involving a population of at-risk, low-socioeconomic status, first-time mothers enrolled in an early intervention home visitation program, Every Child Succeeds (ECS). ECS home visitors from 9 agencies will be randomly assigned to utilize either a specially-designed children's book (intervention) or standard brochures (control) for safe sleep education. Our target enrollment is 230 mothers. Trained ECS home visitors will obtain consent, distribute the book or brochures, and perform baseline assessment of health literacy (via the REALM-R screen), safe sleep knowledge, and home literacy orientation during a third trimester, prenatal home visit. Outcomes data will be collected by the same visitor during subsequent home visits at 1 week old, when infant sleep routines are being established, and 2 months old, at onset of peak SIDS risk. At each visit, the book or brochures will be reviewed.

Outcomes will be compared between intervention and control groups in the following categories: 1) maternal safe sleep knowledge, 2) maternal adherence to safe sleep guidelines (observed), 3) maternal and provider satisfaction with materials utilized to convey safe sleep guidelines, and 4) the degree to which utilizing a children's book for health education impacts home literacy orientation (i.e. attitudes towards reading).

ELIGIBILITY:
Inclusion Criteria:

* Prenatal enrollment in the Every Child Succeeds home visitation program,
* English speaking (intervention book was not available in Spanish), and
* at least 15 years old.

Exclusion Criteria:

* Non-English speaking,
* age under 15 years,
* delayed hospital discharge such that an initial postnatal home visit prior to 3 weeks old is not possible.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change In Maternal Safe Sleep Knowledge | Prenatal baseline to 1 week and 2 months postnatally
  Change in maternal knowledge of safe sleep recommendations (per American Academy of Pediatrics) from a baseline collected prenatally, to outcomes measured at approximately 1 week and then 2 months postnatally.
Assessment of Infant Sleep Environment | During study home visits 1 week and 2 months postnatally
  Direct assessment in the home of infant sleep environment and maternal adherence to American Academy of Pediatrics safe sleep recommendations via the home visitor at approximately 1 week and then 2 months postnatally
Maternal Impression of Safe Sleep Materials Provided | At study home visits 1 week and 2 months postnatally
  Maternal impression of printed materials (book or brochures) used for safe sleep teaching, content and usefulness.
Home Visitor Impression of Safe Sleep Materials Provided | At each study home visit: prenatal, 1 week, and 2 months postnatally
  Home visitor impression of printed materials (book or brochures) used for safe sleep teaching, time of delivery and usefulness.

SECONDARY OUTCOMES:
Maternal Health Literacy Screen | One time prenatally
  Maternal health literacy screen using the validated REALM-R measure (recognizing and pronouncing medical words)
Change in Home Literacy Orientation | Baseline prenatally and 2 months postnatally
  Change is assessed via six questions concerning planned or current shared reading frequency, children's books in the home, and attitudes towards shared reading, as well as attitudes towards and frequency of television use.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Moon RY, Fu L. Sudden infant death syndrome: an update. Pediatr Rev. 2012 Jul;33(7):314-20. doi: 10.1542/pir.33-7-314. PMID 22753789
- [Background] Reich SM, Penner EK, Duncan GJ. Using baby books to increase new mothers' safety practices. Acad Pediatr. 2011 Jan-Feb;11(1):34-43. doi: 10.1016/j.acap.2010.12.006. PMID 21272822
- [Background] Zuckerman B, Khandekar A. Reach Out and Read: evidence based approach to promoting early child development. Curr Opin Pediatr. 2010 Aug;22(4):539-44. doi: 10.1097/MOP.0b013e32833a4673. PMID 20601887
- [Background] Vennemann MM, Hense HW, Bajanowski T, Blair PS, Complojer C, Moon RY, Kiechl-Kohlendorfer U. Bed sharing and the risk of sudden infant death syndrome: can we resolve the debate? J Pediatr. 2012 Jan;160(1):44-8.e2. doi: 10.1016/j.jpeds.2011.06.052. Epub 2011 Aug 24. PMID 21868032
- [Background] Murphy SL, Xu J, Kochanek KD. Deaths: final data for 2010. Natl Vital Stat Rep. 2013 May 8;61(4):1-117. PMID 24979972
- [Background] Wymyslo T, Director. Ohio Child Fatality Review Twelfth Annual Report: 2006-2010, 2012.
- [Background] Maseru, N. P. D., MPH. (2011). Cincinnati-Hamilton County Fetal-Infant Mortality Review. Cincinnat, OH.
- [Background] MacDorman MF, Cnattingius S, Hoffman HJ, Kramer MS, Haglund B. Sudden infant death syndrome and smoking in the United States and Sweden. Am J Epidemiol. 1997 Aug 1;146(3):249-57. doi: 10.1093/oxfordjournals.aje.a009260. PMID 9247009
- [Background] Hauck FR, Thompson JM, Tanabe KO, Moon RY, Vennemann MM. Breastfeeding and reduced risk of sudden infant death syndrome: a meta-analysis. Pediatrics. 2011 Jul;128(1):103-10. doi: 10.1542/peds.2010-3000. Epub 2011 Jun 13. PMID 21669892
- [Background] Moon RY, Tanabe KO, Yang DC, Young HA, Hauck FR. Pacifier use and SIDS: evidence for a consistently reduced risk. Matern Child Health J. 2012 Apr;16(3):609-14. doi: 10.1007/s10995-011-0793-x. PMID 21505778
- [Background] Moon RY, Oden RP, Grady KC. Back to Sleep: an educational intervention with women, infants, and children program clients. Pediatrics. 2004 Mar;113(3 Pt 1):542-7. doi: 10.1542/peds.113.3.542. PMID 14993547
- [Background] Fu LY, Colson ER, Corwin MJ, Moon RY. Infant sleep location: associated maternal and infant characteristics with sudden infant death syndrome prevention recommendations. J Pediatr. 2008 Oct;153(4):503-8. doi: 10.1016/j.jpeds.2008.05.004. Epub 2008 Jun 25. PMID 18582898
- [Background] Robida D, Moon RY. Factors influencing infant sleep position: decisions do not differ by SES in African-American families. Arch Dis Child. 2012 Oct;97(10):900-5. doi: 10.1136/archdischild-2011-301360. Epub 2012 Aug 17. PMID 22904266
- [Background] Ottolini MC, Davis BE, Patel K, Sachs HC, Gershon NB, Moon RY. Prone infant sleeping despite the "Back to Sleep" campaign. Arch Pediatr Adolesc Med. 1999 May;153(5):512-7. doi: 10.1001/archpedi.153.5.512. PMID 10323633
- [Background] Cowan S, Pease A, Bennett S. Usage and impact of an online education tool for preventing sudden unexpected death in infancy. J Paediatr Child Health. 2013 Mar;49(3):228-32. doi: 10.1111/jpc.12128. Epub 2013 Feb 26. PMID 23437780
- [Background] Moult B, Franck LS, Brady H. Ensuring quality information for patients: development and preliminary validation of a new instrument to improve the quality of written health care information. Health Expect. 2004 Jun;7(2):165-75. doi: 10.1111/j.1369-7625.2004.00273.x. PMID 15117391
- [Background] Glascoe FP, Oberklaid F, Dworkin PH, Trimm F. Brief approaches to educating patients and parents in primary care. Pediatrics. 1998 Jun;101(6):E10. doi: 10.1542/peds.101.6.e10. PMID 9606252
- [Background] Barr RG, Rivara FP, Barr M, Cummings P, Taylor J, Lengua LJ, Meredith-Benitz E. Effectiveness of educational materials designed to change knowledge and behaviors regarding crying and shaken-baby syndrome in mothers of newborns: a randomized, controlled trial. Pediatrics. 2009 Mar;123(3):972-80. doi: 10.1542/peds.2008-0908. PMID 19255028
- [Background] Wilson FL, Brown DL, Stephens-Ferris M. Can easy-to-read immunization information increase knowledge in urban low-income mothers? J Pediatr Nurs. 2006 Feb;21(1):4-12. doi: 10.1016/j.pedn.2005.06.003. PMID 16428009
- [Background] Swartz EN. The readability of paediatric patient information materials: Are families satisfied with our handouts and brochures? Paediatr Child Health. 2010 Oct;15(8):509-13. doi: 10.1093/pch/15.8.509. PMID 21966236
- [Background] Dias MS, Smith K, DeGuehery K, Mazur P, Li V, Shaffer ML. Preventing abusive head trauma among infants and young children: a hospital-based, parent education program. Pediatrics. 2005 Apr;115(4):e470-7. doi: 10.1542/peds.2004-1896. PMID 15805350
- [Background] Powell EC, Tanz RR, Uyeda A, Gaffney MB, Sheehan KM. Injury prevention education using pictorial information. Pediatrics. 2000 Jan;105(1):e16. doi: 10.1542/peds.105.1.e16. PMID 10617753
- [Background] NICHD. Safe to Sleep Campaign. 1994-present.; http://www.nichd.nih.gov/sts/Pages/default.aspx.
- [Background] Moon RY, Omron R. Determinants of infant sleep position in an urban population. Clin Pediatr (Phila). 2002 Oct;41(8):569-73. doi: 10.1177/000992280204100803. PMID 12403373
- [Background] Joyner BL, Gill-Bailey C, Moon RY. Infant sleep environments depicted in magazines targeted to women of childbearing age. Pediatrics. 2009 Sep;124(3):e416-22. doi: 10.1542/peds.2008-3735. Epub 2009 Aug 17. PMID 19706591
- [Background] Schuster MA, Duan N, Regalado M, Klein DJ. Anticipatory guidance: what information do parents receive? What information do they want? Arch Pediatr Adolesc Med. 2000 Dec;154(12):1191-8. doi: 10.1001/archpedi.154.12.1191. PMID 11115301
- [Background] National Institutes of Health. Clear Communication: A NIH Health Literacy Initiative. 2013; http://www.nih.gov/clearcommunication/healthliteracy.
- [Background] Yin HS, Johnson M, Mendelsohn AL, Abrams MA, Sanders LM, Dreyer BP. The health literacy of parents in the United States: a nationally representative study. Pediatrics. 2009 Nov;124 Suppl 3:S289-98. doi: 10.1542/peds.2009-1162E. PMID 19861483
- [Background] Sanders LM, Federico S, Klass P, Abrams MA, Dreyer B. Literacy and child health: a systematic review. Arch Pediatr Adolesc Med. 2009 Feb;163(2):131-40. doi: 10.1001/archpediatrics.2008.539. PMID 19188645
- [Background] DeWalt DA, Dilling MH, Rosenthal MS, Pignone MP. Low parental literacy is associated with worse asthma care measures in children. Ambul Pediatr. 2007 Jan-Feb;7(1):25-31. doi: 10.1016/j.ambp.2006.10.001. PMID 17261479
- [Background] Ross LA, Frier BM, Kelnar CJ, Deary IJ. Child and parental mental ability and glycaemic control in children with Type 1 diabetes. Diabet Med. 2001 May;18(5):364-9. doi: 10.1046/j.1464-5491.2001.00468.x. PMID 11472446
- [Background] Morrison AK, Chanmugathas R, Schapira MM, Gorelick MH, Hoffmann RG, Brousseau DC. Caregiver low health literacy and nonurgent use of the pediatric emergency department for febrile illness. Acad Pediatr. 2014 Sep-Oct;14(5):505-9. doi: 10.1016/j.acap.2014.05.001. Epub 2014 Jun 16. PMID 24942934
- [Background] Driessnack M, Chung S, Perkhounkova E, Hein M. Using the "Newest Vital Sign" to assess health literacy in children. J Pediatr Health Care. 2014 Mar-Apr;28(2):165-71. doi: 10.1016/j.pedhc.2013.05.005. Epub 2013 Jul 30. PMID 23910945
- [Background] Abrams MA, Klass P, Dreyer BP. Health literacy and children: recommendations for action. Pediatrics. 2009 Nov;124 Suppl 3:S327-31. doi: 10.1542/peds.2009-1162I. No abstract available. PMID 19861487
- [Background] Davis TC, Mayeaux EJ, Fredrickson D, Bocchini JA Jr, Jackson RH, Murphy PW. Reading ability of parents compared with reading level of pediatric patient education materials. Pediatrics. 1994 Mar;93(3):460-8. PMID 8115206
- [Background] Mendelsohn AL, Mogilner LN, Dreyer BP, Forman JA, Weinstein SC, Broderick M, Cheng KJ, Magloire T, Moore T, Napier C. The impact of a clinic-based literacy intervention on language development in inner-city preschool children. Pediatrics. 2001 Jan;107(1):130-4. doi: 10.1542/peds.107.1.130. PMID 11134446
- [Background] Needlman R, Toker KH, Dreyer BP, Klass P, Mendelsohn AL. Effectiveness of a primary care intervention to support reading aloud: a multicenter evaluation. Ambul Pediatr. 2005 Jul-Aug;5(4):209-15. doi: 10.1367/A04-110R.1. PMID 16026185
- [Background] Sharif I, Rieber S, Ozuah PO. Exposure to Reach Out and Read and vocabulary outcomes in inner city preschoolers. J Natl Med Assoc. 2002 Mar;94(3):171-7. PMID 11918387
- [Background] Berkule SB, Dreyer BP, Huberman HS, Fierman AH, Mendelsohn AL. Attitudes about shared reading among at-risk mothers of newborn babies. Ambul Pediatr. 2007 Jan-Feb;7(1):45-50. doi: 10.1016/j.ambp.2006.10.004. PMID 17261482
- [Background] Berkule SB, Dreyer BP, Klass PE, Huberman HS, Yin HS, Mendelsohn AL. Mothers' expectations for shared reading after delivery: implications for reading activities at 6 months. Ambul Pediatr. 2008 May-Jun;8(3):169-74. doi: 10.1016/j.ambp.2008.01.002. Epub 2008 Apr 8. PMID 18501863
- [Background] Moon RY, Cheng TL, Patel KM, Baumhaft K, Scheidt PC. Parental literacy level and understanding of medical information. Pediatrics. 1998 Aug;102(2):e25. doi: 10.1542/peds.102.2.e25. PMID 9685471
- [Background] Freda MC. The readability of American Academy of Pediatrics patient education brochures. J Pediatr Health Care. 2005 May-Jun;19(3):151-6. doi: 10.1016/j.pedhc.2005.01.013. PMID 15867830
- [Background] Rankin SH, Stallings KD. Patient Education: Principles and Practices. 4th ed. Philadelphia: Lippincott WIlliams and Wilkins; 2001.
- [Background] D'Alessandro DM, Kingsley P, Johnson-West J. The readability of pediatric patient education materials on the World Wide Web. Arch Pediatr Adolesc Med. 2001 Jul;155(7):807-12. doi: 10.1001/archpedi.155.7.807. PMID 11434848
- [Background] Yin HS, Dreyer BP, van Schaick L, Foltin GL, Dinglas C, Mendelsohn AL. Randomized controlled trial of a pictogram-based intervention to reduce liquid medication dosing errors and improve adherence among caregivers of young children. Arch Pediatr Adolesc Med. 2008 Sep;162(9):814-22. doi: 10.1001/archpedi.162.9.814. PMID 18762597
- [Background] French GM, Nicholson L, Skybo T, Klein EG, Schwirian PM, Murray-Johnson L, Sternstein A, Eneli I, Boettner B, Groner JA. An evaluation of mother-centered anticipatory guidance to reduce obesogenic infant feeding behaviors. Pediatrics. 2012 Sep;130(3):e507-17. doi: 10.1542/peds.2011-3027. Epub 2012 Aug 13. PMID 22891225
- [Background] Miller TR, Galbraith M. Injury prevention counseling by pediatricians: a benefit-cost comparison. Pediatrics. 1995 Jul;96(1 Pt 1):1-4. PMID 7596695
- [Background] Muthusamy AD, Leuthner S, Gaebler-Uhing C, Hoffmann RG, Li SH, Basir MA. Supplemental written information improves prenatal counseling: a randomized trial. Pediatrics. 2012 May;129(5):e1269-74. doi: 10.1542/peds.2011-1702. Epub 2012 Apr 9. PMID 22492766
- [Background] Sanders LM, Shaw JS, Guez G, Baur C, Rudd R. Health literacy and child health promotion: implications for research, clinical care, and public policy. Pediatrics. 2009 Nov;124 Suppl 3:S306-14. doi: 10.1542/peds.2009-1162G. PMID 19861485
- [Background] Zuckerman B, Augustyn M. Books and reading: evidence-based standard of care whose time has come. Acad Pediatr. 2011 Jan-Feb;11(1):11-7. doi: 10.1016/j.acap.2010.09.007. PMID 21272819
- [Background] Reich SM, Penner EK, Duncan GJ, Auger A. Using baby books to change new mothers' attitudes about corporal punishment. Child Abuse Negl. 2012 Feb;36(2):108-17. doi: 10.1016/j.chiabu.2011.09.017. Epub 2012 Mar 3. PMID 22391417
- [Background] Bauer NS, Hus AM, Sullivan PD, Szczepaniak D, Carroll AE, Downs SM. A pilot study using children's books to understand caregiver perceptions of parenting practices. J Dev Behav Pediatr. 2012 Jun;33(5):423-30. doi: 10.1097/DBP.0b013e3182560d87. PMID 22495054
- [Background] Reich SM, Bickman L, Saville BR, Alvarez J. The effectiveness of baby books for providing pediatric anticipatory guidance to new mothers. Pediatrics. 2010 May;125(5):997-1002. doi: 10.1542/peds.2009-2728. Epub 2010 Apr 12. PMID 20385630
- [Background] Klass P, Dreyer BP, Mendelsohn AL. Reach out and read: literacy promotion in pediatric primary care. Adv Pediatr. 2009;56:11-27. doi: 10.1016/j.yapd.2009.08.009. No abstract available. PMID 19968940
- [Background] Hartling L, Scott S, Pandya R, Johnson D, Bishop T, Klassen TP. Storytelling as a communication tool for health consumers: development of an intervention for parents of children with croup. Stories to communicate health information. BMC Pediatr. 2010 Sep 2;10:64. doi: 10.1186/1471-2431-10-64. PMID 20813044
- [Background] Surber J. Effect of topic label repetition and importance on reading time and recall of text. J Educ Psychology. 2001;93(2):279-287.
- [Background] Nyhout A, O'Neill D. Mothers' complex talk when sharing books with their toddlers: book genre matters. First Language. 2013;33(2):115-131.
- [Background] Every Child Succeeds. 2013; http://www.everychildsucceeds.org/Our-Mission.aspx.
- [Background] Davis TC, Long SW, Jackson RH, Mayeaux EJ, George RB, Murphy PW, Crouch MA. Rapid estimate of adult literacy in medicine: a shortened screening instrument. Fam Med. 1993 Jun;25(6):391-5. PMID 8349060
- [Background] Bass PF 3rd, Wilson JF, Griffith CH. A shortened instrument for literacy screening. J Gen Intern Med. 2003 Dec;18(12):1036-8. doi: 10.1111/j.1525-1497.2003.10651.x. PMID 14687263
- [Background] Task Force on Sudden Infant Death Syndrome; Moon RY. SIDS and other sleep-related infant deaths: expansion of recommendations for a safe infant sleeping environment. Pediatrics. 2011 Nov;128(5):1030-9. doi: 10.1542/peds.2011-2284. Epub 2011 Oct 17. PMID 22007004
- [Background] Hutton JS, Busch L. Sleep Baby, Safe and Snug. Cincinnati, OH: blue manatee press; 2013.
- [Background] Whitehurst GJ. Dialogic Reading: An Effective Way to Read to Preschoolers. 2013; http://www.readingrockets.org/article/400/.
- [Background] Council on Communications and Media; Brown A. Media use by children younger than 2 years. Pediatrics. 2011 Nov;128(5):1040-5. doi: 10.1542/peds.2011-1753. Epub 2011 Oct 17. PMID 22007002
- [Background] Duch H, Fisher EM, Ensari I, Harrington A. Screen time use in children under 3 years old: a systematic review of correlates. Int J Behav Nutr Phys Act. 2013 Aug 23;10:102. doi: 10.1186/1479-5868-10-102. PMID 23967799
- [Background] Mendelsohn AL, Berkule SB, Tomopoulos S, Tamis-LeMonda CS, Huberman HS, Alvir J, Dreyer BP. Infant television and video exposure associated with limited parent-child verbal interactions in low socioeconomic status households. Arch Pediatr Adolesc Med. 2008 May;162(5):411-7. doi: 10.1001/archpedi.162.5.411. PMID 18458186
- [Derived] Hutton JS, Lin L, Gruber R, Berndsen J, DeWitt T, Van Ginkel JB, Ammerman RT. Shared Reading and Television Across the Perinatal Period in Low-SES Households. Clin Pediatr (Phila). 2018 Jul;57(8):904-912. doi: 10.1177/0009922817737077. Epub 2017 Oct 25. PMID 29067842